CLINICAL TRIAL: NCT03303404
Title: 24-hour Blood Pressure Measurements and Ischemic Conditioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-07-0043
Record Dates: First submitted 2017-10-02; First posted 2017-10-06 (Actual); Results first posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Blood Pressure
MeSH Terms: interventions — Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Ambulatory (24-hour) Blood Pressure (Experimental)
  Interventions: Device: Ambulatory (24-hour) Blood Pressure

INTERVENTIONS:
Device: Ambulatory (24-hour) Blood Pressure — Unlike casual blood pressure measurements, 24-hour ambulatory blood pressure monitoring provides an insight into blood pressure changes in everyday life and an estimate of the overall blood pressure load exerted on the cardiovascular system over 24 hours. Blood pressure recordings over a 24-hour period of normal daily activity will be made using a noninvasive ambulatory monitor (Spacelabs, Redlands, WA). The ambulatory system will be calibrated against a mercury sphygmomanometer, and the cuff will be programmed to inflate automatically every 15 min from 6 AM to 11 PM and every 20 min between 11 PM and 6 AM. For each individual subject, the nighttime period will be defined as the time when the subject goes to bed at night until rising in the morning. Daytime will be defined as the remainder of the 24-hour period. Daytime and nighttime states will be monitored by an Actiwatch (Mini-MItter, Bend, OR), a watch-like device placed on the wrist that measures gross motor activity.

SUMMARY:
To determine if 24-hr ambulatory blood pressure monitoring effects endothelial function, we will measure flow-mediated dilation before and after the blood pressure monitoring (ischemia conditioning).

DETAILED DESCRIPTION:
Reestablishing blood flow (reperfusion) to organs that had their blood supply restricted (ischemia) can cause damage to the vasculature via injury and tissue death resulting in endothelial dysfunction. This ischemia-reperfusion (blood flow occlusion and resupply) triggered injury can be reduced or prevented by preceding brief periods of ischemia called preconditioning. Properly-performed preconditioning can exert a powerful protection against a subsequent sustained period of ischemia in a variety of organs in the body including the heart, kidney, and skeletal muscle. Preconditioning protocol involves repeated brief inflation and deflation of a blood pressure cuff. In many of human cardiovascular research studies, it is common to measure endothelial function and ambulatory (24-hour) blood pressure. The ambulatory blood pressure device takes repeated blood pressure readings every 15-30 minutes during the daytime and 30-60 minutes at night. It is possible that repeated bouts of inflation/deflation of the blood pressure cuff could induce preconditioning effects and influence endothelial function. Therefore, in the proposed study we aim to address this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

Adults aged between 30 to 60 years old.

Exclusion Criteria:

Exclusion from the study may be due to: i) pregnancy (by asking the subjects when the last time she had menstruation; we do have simple testing kits available if a subject is unsure about her status); ii) a recent illness, recent surgery, or any medical intervention in the 48 hours before any of the study days; iii) personal history of diabetes (fasting blood glucose > 126 mg/dL), heart disease, or other cardiovascular problems.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Hirofumi Tanaka, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fico BG, Zhu W, Tanaka H. Does 24-h ambulatory blood pressure monitoring act as ischemic preconditioning and influence endothelial function? J Hum Hypertens. 2019 Nov;33(11):817-820. doi: 10.1038/s41371-019-0214-y. Epub 2019 Jun 27. PMID 31249371

RESULTS

PARTICIPANT FLOW:
Groups:
- Ambulatory (24-hour) Blood Pressure: Ambulatory (24-hour) Blood Pressure: Unlike casual blood pressure measurements, 24-hour ambulatory blood pressure monitoring provides an insight into blood pressure changes in everyday life and an estimate of the overall blood pressure load exerted on the cardiovascular system over 24 hours. Blood pressure recordings over a 24-hour period of normal daily activity will be made using a noninvasive ambulatory monitor (Spacelabs, Redlands, WA). The ambulatory system will be calibrated against a mercury sphygmomanometer, and the cuff will be programmed to inflate automatically every 15 min from 6 AM to 11 PM and every 20 min between 11 PM and 6 AM. For each individual subject, the nighttime period will be defined as the time when the subject goes to bed at night until rising in the morning. Daytime will be defined as the remainder of the 24-hour period.
Period: Overall Study
Arm/Group | Ambulatory (24-hour) Blood Pressure
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ambulatory (24-hour) Blood Pressure
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Flow Mediated Dilation After 24 Hour Ischemic Conditioning With Blood Pressure Cuff
Description: Flow-mediated dilatation (FMD) is a common and non-invasive method to assess vascular endothelial function by measuring the Brachial artery's responsiveness (diameter percent increase) following a brief period of occlusion.
Time Frame: Baseline, Post 24 hour conditioning
Measure: Mean (Standard Deviation); unit: percentage of baseline
Groups:
- Intervention: This is a single arm acute intervention study.
Arm/Group | Intervention
Number analyzed (Participants) | 22
percentage of baseline | 6.6 (2.0)

ADVERSE EVENTS:
Time Frame: 6 months
Description: The procedures to be used in this investigation posed very minimal risk to our subjects.
Groups:
- Intervention: This is a single arm study did not involve grouping.
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT03303404/Prot_SAP_000.pdf